CLINICAL TRIAL: NCT07357727
Title: A Phase 3, Randomized, Double-blind, Active-control Study of Pelabresib (DAK539) and Ruxolitinib vs. Placebo and Ruxolitinib in Adult Patients With Myelofibrosis Who Are JAK Inhibitor Naive
Brief Title: A Phase 3 Study of Pelabresib (DAK539) and Ruxolitinib in Myelofibrosis (MF)
Acronym: MANIFEST-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDAK539A12303; 2025-523555-66-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2026-01-15; First posted 2026-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Primary Myelofibrosis (PMF); Post-polycythemia Vera Myelofibrosis (PPV-MF); Post-essential Thrombocythemia Myelofibrosis (PET-MF)
Keywords: Pelabresib (DAK539); Ruxolitinib; Adult participants; Myelofibrosis (MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pelabresib + Ruxolitinib (Experimental): Participants in this arm receive pelabresib (DAK539) orally once daily for 14 days of each 21-day cycle, in combination with ruxolitinib, which is taken orally twice daily throughout each cycle. Participants may continue receiving study treatment until they experience unacceptable toxicity, disease progression, or until either the investigator or the participant decides to discontinue treatment.
  Interventions: Drug: Pelabresib; Drug: Ruxolitinib
- Arm 2: Placebo + Ruxolitinib (Placebo Comparator): Participants in this arm receive a matching placebo orally once daily for 14 days of each 21-day cycle, together with ruxolitinib, which is also taken orally twice daily throughout each cycle.
  Participants may continue receiving study treatment until they experience unacceptable toxicity, disease progression, or until either the investigator or the participant decides to discontinue treatment.
  Interventions: Drug: Ruxolitinib; Drug: Placebo

INTERVENTIONS:
Drug: Pelabresib — Pelabresib monohydrate tablets
  Other Names: DAK539
  Arms: Arm 1: Pelabresib + Ruxolitinib
Drug: Ruxolitinib — Ruxolitinib phosphate tablets
  Other Names: INC424
Drug: Placebo — Matches pelabresib
  Arms: Arm 2: Placebo + Ruxolitinib

SUMMARY:
The purpose of this trial is to evaluate whether treatment with pelabresib in combination with ruxolitinib leads to improved clinical outcomes compared to ruxolitinib alone in patients with primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PPV-MF), or post-essential thrombocythemia myelofibrosis (PET-MF) who have not previously received Janus kinase (JAK) inhibitor therapy.

DETAILED DESCRIPTION:
The study for each participant is composed of several distinct periods: a screening period, a study treatment period, and a post-treatment follow-up phase.

1. Screening Period:

   The screening period lasts for up to 28 days prior to Cycle 1 Day 1, which marks the beginning of treatment. During this time, the participant's eligibility for the study is confirmed, informed consent is obtained, and all required baseline assessments are completed.
2. Treatment Period:

   The treatment period begins on Cycle 1 Day 1, which is the point of randomization and the start of study treatment. This period continues until the participant permanently discontinues study treatment, which may occur due to disease progression, unacceptable toxicity, participant withdrawal, or other reasons specified in the protocol. Throughout this period, participants receive study drugs in 21-day cycles, with pelabresib or placebo administered for 14 days and ruxolitinib given continuously. Regular site visits and assessments are conducted according to the Schedule of Activities.
3. Safety Follow-up Period:

   The safety follow-up period extends for 30 days (with a window of plus or minus 3 days) after the participant receives their last dose of pelabresib or placebo. During this period, participants are monitored for any late-onset adverse events or safety concerns that may arise after discontinuing the study treatment.
4. Efficacy Follow-up Period:

   Following the safety follow-up, efficacy follow-up visits are scheduled every 12 weeks for participants who have not shown evidence of disease progression, meaning there is no documented progression of splenomegaly or leukemic transformation and no new therapy for myelofibrosis has been started. The purpose of this follow-up is to continue monitoring efficacy endpoints, such as spleen imaging, laboratory assessments, and bone marrow biopsies, until either disease progression occurs or a new therapy is initiated.
5. Survival Follow-up Period:

Once a participant enters the survival follow-up phase, follow-up visits are conducted every 12 weeks and may be performed remotely. This phase applies to participants who have experienced documented disease progression or have started a new therapy for myelofibrosis. The aim of survival follow-up is to monitor overall survival and to collect ongoing data regarding disease status and any subsequent therapies the participant may receive.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants have diagnosis of primary myelofibrosis (PMF) or post-polycythemia vera myelofibrosis (post-PV MF) or post-essential thrombocythemia myelofibrosis (post-ET MF) according to the International Consensus Classification (ICC) of Myeloid Neoplasms and Acute Leukemias 2022
* DIPSS risk category of intermediate-1, intermediate-2 or high-risk
* Spleen volume ≥ 450 cm3 by CT or MRI scan (local read sufficient if no central read available)
* Have an average TSS of ≥15 within 7 days prior to randomization, using MFSAF v. 4.0 (at least 4 out of 7 TSS assessments required for average calculation)
* Participants with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Blasts <5% in peripheral blood. Assessment of blasts in peripheral blood is mandatory at screening
* Platelet count ≥ 100 x 10^9/L in the absence of growth factors or transfusions for the previous 4 weeks

Key Exclusion Criteria:

* Prior splenectomy at any time or splenic irradiation in the previous 6 months
* Prior hematopoietic cell transplant or participant anticipated to receive a hematopoietic cell transplant within 24 weeks from the date of randomization
* Blasts ≥ 5% in bone marrow if results available at screening or history of accelerated phase (AP) or leukemic transformation
* History of a malignancy (other than MF, PPV-MF or PET-MF) in the past 3 years in need of systemic treatment
* Received any approved or investigational agent other than hydroxyurea or anagrelide for the treatment of MF within 14 days of first dose of study treatment or within 5 half-lives of the approved or investigational agent, whichever is longer
* Prior treatment with any JAK inhibitor or Bromodomain and extraterminal domain (BET) inhibitor

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2028-05-17 (Estimated); Study Completion 2030-12-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Splenic Response (SVR35) by Central Radiology Reads at Week 24 in participants with baseline total symptom score (TSS) ≥ 25 | Week 24
  Spleen Response (SVR35) is defined as achieving a reduction of at least 35 percent in spleen volume from baseline to Week 24, as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and assessed by a centralized radiology review in participants with baseline TSS ≥ 25.
Absolute change from baseline in total symptom score (TSS) at Week 24 in participants with baseline TSS ≥ 25 | Baseline, Week 24
  Symptom improvement at Week 24 is defined as the absolute change from baseline in the total symptom score (TSS) at Week 24, as measured by the Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0) in participants with baseline TSS ≥ 25.
Number of Participants with Splenic Response (SVR35) by Central Radiology Reads at Week 24 in participants with baseline TSS ≥ 15 | Week 24
  Spleen Response (SVR35) is defined as achieving a reduction of at least 35 percent in spleen volume from baseline to Week 24, as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and assessed by a centralized radiology review in participants with baseline TSS ≥ 15.
Absolute change from baseline in total symptom score (TSS) at Week 24 in participants with baseline TSS ≥ 15 | Baseline, Week 24
  Symptom improvement at Week 24 is defined as the absolute change from baseline in the total symptom score (TSS) at Week 24, as measured by the Myelofibrosis Symptom Assessment Form version 4.0 (MFSAF v4.0) in participants with baseline TSS ≥ 15.

SECONDARY OUTCOMES:
Number of Participants with Splenic Response (SVR35) by Central Radiology Reads over time | Week 12, Week 36, Week 48 and every 12 weeks thereafter till End of Study (an average of 3 years)
  Spleen Response (SVR35) over time is defined as achieving a reduction of at least 35 percent in spleen volume from baseline to Week 12, Week 36, Week 48 and thereafter, as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and assessed by a centralized radiology review.
Absolute change from baseline and percentage change from baseline in spleen volume over time | Baseline, Week 12, Week 24, Week 36, Week 48, and every 12 weeks thereafter till End of Study (an average of 3 years)
  Absolute and percentage change from baseline in spleen volume over time will be summarized using descriptive summary statistics
Time to first SVR35 response | From date of randomization to the date of first SVR35 response, assessed up to approximately 3 years
  Time to first SVR35 response defined as the time from date of randomization to the date of first SVR35 response as measured by MRI (or CT scan) will be summarized by treatment arm.
Duration of first SVR35 response | From first SVR35 response to loss of response, assessed up to approximately 3 years
  Duration of first SVR35 response defined as the time from first SVR35 response to loss of response for any participant who reaches SVR35 at any time.
Number of Participants with TSS50 response at Week 24 | Week 24
  Symptom response defined as achieving ≥ 50% reduction in total symptom score (TSS50) from baseline to Week 24 as measured by the MFSAF v4.0
Number of Participants with TSS50 response over time | Baseline, Week 12, Week 24, Week 36, Week 48, and every 12 weeks thereafter till End of Study (an average of 3 years)
  Symptom response defined as achieving ≥ 50% reduction in total symptom score (TSS50) from baseline to Week 12, Week 36, Week 48 and thereafter as measured by the MFSAF v4.0
Absolute and percentage change from baseline in TSS over time | Baseline, Week 12, Week 24, Week 36, Week 48, and every 12 weeks thereafter till End of Study (an average of 3 years)
  Absolute change from baseline and percentage change from baseline in TSS over time
Time to first TSS50 response | From date of randomization till date of first TSS50 response, assessed up to approximately 3 years
  Time to first TSS50 response defined as the time from date of randomization to the date of first TSS50 response as measured by the MFSAF v4.0.
Duration of TSS50 response | From first TSS50 response to loss of response, assessed up to approximately 3 years
  Duration of TSS50 response defined as the time from first TSS50 response to loss of response for any participant who reaches TSS50 at any time.
Dual Response (SVR35 + TSS50) | Baseline, Week 12, Week 24, Week 36, Week 48, and every 12 weeks thereafter till End of Study (an average of 3 years)
  Dual response is defined as achieving both ≥ 35% reduction in spleen volume (SVR35) and ≥ 50% reduction in total symptom score (TSS50) from baseline to Week 12, 24, 36, 48 and every 12 weeks thereafter, with SVR measured by MRI (or CT scan) and assessed by central radiology read and TSS measured by MFSAF v4.0.
Hemoglobin response | 12 consecutive weeks (rolling window) up to 7 days following last dose of pelabresib/placebo
  Hemoglobin response defined as a ≥1.5 g/dL average increase in hemoglobin from baseline in any 12-week mean hemoglobin concentration.
Change from baseline in hemoglobin over time | Up to 7 days following last dose of pelabresib/placebo
  Change from baseline in hemoglobin over time will be summarized using descriptive summary statistics.
Anemia response over time | Up to 7 days following last dose of pelabresib/placebo
  Anemia response (major response, minor response, stable anemia, progressive anemia) as per proposed 2024 IWG-ELN criteria in participants with transfusion dependent and non-transfusion dependent anemia (Tefferi et al 2024).
Overall survival (OS) | From date of randomization till date of death due to any cause, assessed up to approximately 3 years
  Overall survival (OS) defined as the time from date of randomization to date of death due to any cause.
Progression-free survival (PFS) | From date of randomization till date of documented disease progression, or death due to any cause whichever comes first, assessed up to approximately 3 years
  Progression-free survival (PFS) defined as the time from date of randomization to date of documented disease progression, or death due to any cause whichever comes first.
Leukemia-free survival (LFS) | From date of randomization till date of leukemic transformation, or death due to any cause whichever comes first, assessed up to approximately 3 years
  Leukemia-free survival (LFS) is defined as the time from date of randomization to date of leukemic transformation, or death due to any cause whichever comes first.
Exposure-Adjusted Incidence Rate (EAIR) of Participants with Leukemic Transformation | Throughout study completion (an average of 3 years)
  The EAIR of participants with leukemic transformation is the rate at which this event occurs, adjusted for the actual time participants were exposed to the study drug(s).
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days following last dose of pelabresib/placebo
  Incidence of adverse events by type, frequency, and severity, as graded by the NCI CTCAE version 5.0.
Pelabresib plasma concentrations | Cycle 1: Day 1 (0/Pre-dose and 0.5 post dose), Day 7 (0/Pre-dose), Day 14 (0/Pre-dose, 2, and 5 hours post-dose). 1 cycle = 21 days.
  Blood samples for pelabresib pharmacokinetics (PK) will be obtained and evaluated in all participants at all dose levels and summarized using descriptive statistics.
Maximum observed plasma Concentration (Cmax) of pelabresib in participants enrolled in China and Japan | Cycle 1 Day Day 14 (0/Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose). 1 cycle = 21 days.
  Venous whole blood samples will be collected for pharmacokinetic characterization in a subset of participants enrolled in China and Japan. Cmax will be listed and summarized using descriptive statistics.
Time to Maximum observed plasma Concentration (Tmax) of pelabresib in participants enrolled in China and Japan | Cycle 1 Day Day 14 (0/Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose). 1 cycle = 21 days.
  Venous whole blood samples will be collected for pharmacokinetic characterization in a subset of participants enrolled in China and Japan. Tmax will be listed and summarized using descriptive statistics.
Area Under the Concentration-Time Curve over a dosing interval (AUCtau) of pelabresib in participants enrolled in China and Japan | Cycle 1 Day Day 14 (0/Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose). 1 cycle = 21 days.
  Venous whole blood samples will be collected for pharmacokinetic characterization in a subset of participants enrolled in China and Japan. AUCtau will be listed and summarized using descriptive statistics.
Change from baseline over time in fatigue as measured by PROMIS SF v1.0 Fatigue 7a | Baseline, once per week from Cycles 1 to 9 (each cycle is 21 days), day 1 of every odd cycle thereafter, within 7 days of last dose of pelabresib/placebo and at 12 weeks following last dose of pelabresib/placebo
  The PROMIS Short Form version 1.0 Fatigue 7a is a seven-question survey that measures how much fatigue has affected a person over the past week. Each question is rated from "Never" to "Always" on a five-point scale. The total score is converted to a standardized score, where the average is 50 and the standard deviation is 10.
  A lower score means less fatigue and minimal impact on daily life, while a higher score indicates more severe fatigue and greater disruption of daily activities.
Change from baseline over time in overall QOL and functional scales as measured by the EORTC QLQ-C30 | Baseline, day 1 of every cycle from Cycle 1 to 9 (each cycle is 21 days), day 1 of every odd cycle thereafter, within 7 days of last dose of pelabresib/placebo and at 12 weeks following last dose of pelabresib/placebo
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) measures overall quality of life and key functional areas in people with cancer, including physical, role, emotional, cognitive, and social functioning.
  Items are rated from 1 (not at all) to 4 (very much), except for the global quality of life scale, which uses a 1 to 7 scale.
  Scores are converted to a 0 to 100 scale.
  Higher scores indicate better functioning and quality of life, while lower scores reflect poorer functioning and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com